CLINICAL TRIAL: NCT07126444
Title: Effects of an Exercise Snack Intervention on Employee Health and Work Performance: A Study at Kaohsiung Medical University
Brief Title: Effects of an Exercise Snack Intervention on Employee Health and Work Performance
Status: Not yet recruiting | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-F(I)-20250189; 113825017999UC003-6 (Other Grant/Funding Number: Kaohsiung Medical University)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: Occupational Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — No biospecimens will be collected in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Employee: Employees of Kaohsiung Medical University, including faculty and administrative staff. Participants are adults (≥20 years) currently working full-time or part-time at the university. This group is selected because prolonged sedentary work and job-related demands are associated with musculoskeletal discomfort, stress, and reduced physical activity. They represent the target population for evaluating the feasibility and effectiveness of brief workplace exercise interventions ("exercise snacks").

SUMMARY:
To create brief exercise videos addressing physical discomfort, fitness goals, and movement skills.

To design personalized exercise menus to enhance staff adherence.

To apply the "exercise snacking" model with multiple short daily sessions and evaluate its effects on health, work performance, and exercise behavior.

DETAILED DESCRIPTION:
1. To develop brief exercise videos targeting different areas of physical discomfort (e.g., neck and shoulders, lower back, lower limbs), specific fitness goals (e.g., localized muscle stretching, targeted muscle strengthening, cardiorespiratory endurance, balance training), high-intensity interval training (HIIT), or the acquisition of specific movement skills (e.g., core stability, pelvic floor muscle contraction, and multi-directional pelvic mobility).
2. To design personalized exercise "menus" based on individual needs identified through a preliminary assessment, with the goal of improving adherence to voluntary exercise routines among staff.
3. To apply the concept of "exercise snacking" by implementing a daily routine of 3 to 8 brief exercise sessions, and to evaluate changes in staff members' physiological health, work performance, and exercise behavior after a 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Currently employed at Kaohsiung Medical University or Kaohsiung Medical University Hospital.
2. Willing to participate in a 12-week exercise intervention, complete related questionnaires, and undergo physical performance assessments.

Exclusion Criteria:

1. Pregnant individuals, due to safety concerns related to exercise intensity and physical assessments.
2. Individuals with a diagnosed neurological disorder (e.g., stroke, Parkinson's disease).
3. Individuals experiencing severe pain in the upper or lower limb joints that interferes with their ability to complete the assessments.
4. Individuals assigned to high-intensity exercise who have unstable cardiac conditions (e.g., angina, myocardial infarction, heart failure).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit full-time faculty and staff from a university and its affiliated hospital. The participants are generally healthy adults who may experience varying levels of musculoskeletal discomfort or reduced physical fitness due to prolonged sedentary or standing work conditions. Individuals are expected to be capable of independent physical activity and willing to engage in brief, self-directed exercise sessions integrated into their daily routine.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-08-29 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical fitness test | 30 minutes
Work Ability Index | 5 minutes
Copenhagen Burnout Inventory | 5 minutes
Perceived Stress Scale-14 | 5 minutes
Exercise adherence | 1 minutes/per day

CONTACTS AND LOCATIONS:
Overall Officials: Lih-Jiun Liaw, Study Chair — Kaohsiung Medical University

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT07126444/Prot_000.pdf